CLINICAL TRIAL: NCT04496999
Title: HDM201 and Midostaurin (HDMM) in Relapsed/Refractory AML With FLT3mut and TP53wt; a Phase I Study.
Brief Title: HDM201 and Midostaurin (HDMM) in Relapsed/Refractory AML With FLT3mut and TP53wt.
Acronym: HDMM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDMM
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: AML, Adult
Keywords: AML with FLT3-ITD or FLT3-TKD and TP53wt; relapsed/refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — siremadlin; midostaurin

STUDY DESIGN:
Intervention Model Description: Non-randomized prospective open-label single-arm clinical phase I trial investigating dose finding, feasibility and safety of the combined treatment of HDM201 and midostaurin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Midostaurin with HDM201 dose escalation. (Experimental): Midostaurin 50mg bid d1-28 (morning, evening) and HDM201
  Interventions: Drug: HDM201; Drug: Midostaurin

INTERVENTIONS:
Drug: HDM201 — Dose level 0: HDM201 40 mg QD d1,2 (midday)/ Dose level 1: HDM201 40 mg QD d1,2,3 (midday) = Starting dose/ Dose level 2: HDM201 40 mg QD d1,2,3,4,5 (midday)/ Dose level 3: HDM201 60 mg QD d1,2,3,4,5 (midday)/ Dose level 4: HDM201 80 mg QD d1,2,3,4,5 (midday)
  Other Names: Dose finding
Drug: Midostaurin — Midostaurin 50mg bid d1-28 (morning, evening)

SUMMARY:
This is a non-randomized prospective open-label single-arm clinical phase I trial investigating dose finding, feasibility and safety of the combined treatment of HDM201 and midostaurin in patients with relapsed/refractory acute myeloid leukemia (AML) with FLT3mut applying an accelerated titration design.

DETAILED DESCRIPTION:
Background and Rationale:

Acute myeloid leukemia (AML) is a clonal hematopoietic malignant disease characterized by genetic and epigenetic alterations leading to inactivation of the tumor suppressor p53. This contributes to a block in normal differentiation of the various blood type lineages and to an accumulation of leukemic blasts in the blood and bone marrow. The disease variants have been grouped into favorable, intermediate and poor risk categories. The largest group of poor risk AML is characterized by the genetic alterations of the FLT3 receptor gene termed FLT3-ITD or FLT3-TKD. The prognosis for this specific subset which comprises 25-35% of all AML patients is generally poor, particularly in elderly or in relapsed patients, highlighting the unmet need for novel treatments.

Targeting the mutated FLT3 receptor is a promising approach to treat this specific poor risk AML subset. Midostaurin is particularly effective to induce cell death in FLT3-ITD/-TKD and TP53wt cells. Targeting MDM2 is a novel approach to restore the crucial p53 tumor suppressor function in AML cells. Preliminary data indicate that the MDM2 inhibitor HDM201 is active in AML cell lines in vitro and in vivo. Like midostaurin HDM201 is specifically effective to induce cell death in FLT3-ITD and TP53wt cells. The combination of midostaurin and HDM201 targets FLT3-ITD AML cells, with little effect on FLT3 wt cells and healthy blood cells. Both compounds induce apoptosis and cell death in a dose-dependent manner in FLT3-ITD TP53wt AML cells, with enhanced effects in the combination treatment. The combination treatment with midostaurin and HDM201 ought to be superior to the current best available treatment which utilizes intensive genotoxic induction therapy. In order to confirm inhibition of mutated FLT3 receptor and restoration of p53 tumor suppressor function, blood samples will be analyzed in this trial before, during and after treatment with HDM201 and midostaurin for changes in the expression of FLT3 and p53 target genes as well as induction of pro- apoptotic genes. These gene expression levels will be correlated with clinical response and outcome.

Objectives:

Primary objective:

The primary objective of this trial is to establish the recommended dose for a subsequent phase II (RP2D) of HDM201 in combination with midostaurin in patients with relapsed or refractory FLT3mut TP53wt AML.

Secondary objectives:

The secondary objectives are to determine the safety and tolerability of HDM201 in combination with midostaurin and to assess the preliminary antitumor activity of HDM201 in combination with midostaurin in patients with relapsed or refractory FLT3mut TP53wt AML and in newly diagnosed AML with FLT3mut and TP53wt.

Study Duration:

The trial study duration encompasses the time from when the first participant signs the informed consent until the last protocol-specific procedure of the last patient in the trial has been completed.

This phase I trial involves a minimum of 3 and a maximum of 24 subjects. Accordingly, the Investigator anticipate a duration of recruitment of between 3 and 18 months.

All patients will be followed up for up to 12 months after end of treatment, adding to a total study duration of between 15 and 33 months depending on the effective number of patients in the various dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

* AML with FLT3-ITD or FLT3-TKD and TP53wt.
* Age over 18 years
* Patient must give written informed consent before registration indicating that the patient understands the purpose of the procedures required for the trial and is willing to participate in the trial.
* Patients with relapsed/refractory disease must have morphologic proof (from bone marrow aspirate, smears or touch preps of bone marrow biopsy) of AML with >= 10% blasts within two weeks (14 days) prior to initiation of therapy.
* Patients must demonstrate one of the following: Relapse after first complete remission or refractory to conventional induction chemotherapy with or without Midostaurin (failure to respond to 1 or more cycles of daunorubicin and cytarabine) or to re-induction.
* Patients with relapse after HSCT (non-preventive) and pretransplant treatment with Midostaurin (FLT3-ITD or FLT3-TKD at diagnosis) or without Midostaurin (acquired FLT3 mutation).
* Laboratory values that indicate adequate organ function assessed locally at the screening visit:

  * AST ≤ 3 times ULN
  * Alanine aminotransferase (ALT) ≤ 3 times ULN
  * Serum total bilirubin ≤ 1.5 times ULN, unless in case of hyperbilirubinemia due to an isolated Gilbert syndrome
  * Estimated (by Cockcroft-Gault) creatinine clearance ≥ 30ml/min
* ECOG score performance status 0-2.
* Patients may have received therapy for other malignancies, as long as they have completed therapy at least 6 months prior to study entry.
* Subjects must have a life expectancy of 3 or more months.

Exclusion Criteria:

* AML with FLT3wt or TP53mut
* Ongoing adverse event drug-induced neuropathy of prior therapy grade ≥2 (according to CTCAE criteria Version 5.0) at registration
* Previous malignancy within 2 years with the exception of adequately treated in situ cervical cancer or localized non-melanoma skin cancer.
* Evidence of ongoing uncontrolled systemic infections.
* Major surgery within 4 weeks prior to trial registration
* Concurrent treatment with other experimental drugs or treatment in a clinical trial within 30 days prior to trial registration.
* Treatment with chemotherapy and radiotherapy within 3 weeks prior to trial registration
* Vaccinated with live, attenuated vaccines within 4 weeks prior to trial registration
* History of stroke or intracranial hemorrhage within 6 months prior to trial registration.
* Clinically significant cardiovascular disease such as congestive heart failure NYHA III or IV (as defined by the New York Heart Association Functional Classification), uncontrolled or symptomatic arrhythmias, unstable angina pectoris, myocardial infarction within 6 months of prior to registration
* Prior solid organ transplantation
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion,

  * could impair the ability of the patient to participate in the trial
  * could compromise the patient's safety,
  * could interfere with the absorption or metabolism of midostaurin or HDM201,
  * could put the trial outcomes at undue risk,
  * could prevent compliance with trial treatment.
* Psychiatric disorder precluding understanding of trial information, giving informed consent, or interfering with compliance for oral drug intake.
* Known hypersensitivity to trial drug(s) or hypersensitivity to any other component of the trial drugs.
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol and follow-up.
* Impairment of gastrointestinal (GI) function or GI disease that might alter significantly the absorption of midostaurin and/or HDM201.
* Known confirmed diagnosis of HIV infection or active viral hepatitis (testing is not mandatory to exclude these viral infections).
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for at least 12 months after stopping medication. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 12 months prior to screening). The vasectomized male partner should be the sole partner for that subject
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
  * Midostaurin may reduce the effectiveness of hormonal contraceptives; therefore, females using systemically active hormonal contraceptives should add a barrier method of contraception.

Women are considered post-menopausal and not of child bearing potential if they have had 2 years of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

* Sexually active males unless they use a condom during intercourse while taking the drug during treatment, and for at least 12 months after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via semen.
* Unwillingness or inability to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Dose finding | 30 days
  to identify the incidence of dose limiting toxicities (DLT) at each dose level and to determine the maximum tolerated dose (MTD) of HDM201 and its recommended dose that will be used in a later phase II study (recommended phase II dose; RP2D) when added to midostaurin

SECONDARY OUTCOMES:
Overall response rate (ORR) | 60 days
  CR, CRi, CRp, PR including assessment of minimal residual disease by molecular diagnostics and flowcytometry after cycles 1 and 2.
Adverse Events | 33 months
  Number of patients experiencing adverse events and severity of the adverse events
Progression free survival | 33 months
  Time from end of treatment (after bone marrow assessment after cycle 2) until progression of disease or death as a result of any cause.
Overall survival | 33 months
  Time from end of treatment (after bone marrow assessment after cycle 2) until death as a result of any cause.
Infectious complications of study treatment | 33 months
  Assessment of the number of febrile episodes requiring antibiotic/antifungal treatment as well as assessment of identified causing germs.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pabst, Prof, Study Chair — Department of Medical Oncology, University Hospital Bern Switzerland
Locations (1):
- Departement of Medical Oncology, University Hospital Berne, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes